CLINICAL TRIAL: NCT04592991
Title: Targeted Molecular Probe for Abdominal Aortic Aneurysm Imaging and Therapy
Brief Title: CCR2 AAA Pilot Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We were only able to enroll 1 subject so we had no way to compare a control or other study groups and develop any kind of results. This study is essentially the same study as NCT04586452, which we would like to place focus and effort on that study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 202004104
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: There will be two (2) groups in this study. We plan to recruit 5 patients with AAA and 3 patients with diagnosed non-aneurysmal (without aneurysm) aortoiliac occlusive disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AAA Group (Active Comparator): Participants with AAA will undergo routine clinical evaluation of AAA including ultrasound and CT and scheduling of open surgical repair as directed by the treating physician. We will record age and tobacco use of participant. If participant has not had a renal function blood test performed within the past 90 days, we will draw approximately 2 teaspoons of blood for a creatinine test. We will also ask the participant's permission to use a contrast dye for the CT portion of the PET-CT scan. If the participant agrees we will additional questions to gauge eligibility to receive the contrast dye.
  If available, we would like to collect any discarded AAA tissue from the surgical procedure. This discarded tissue will be kept as part of a Washington University vascular research repository. If the participant agrees to this there will be a separate consent form to sign allowing the collection of the leftover tissue along with some information about medical history.
  Interventions: Diagnostic Test: AAA Group- PET-CT imaging with injection of 64Cu-DOTA-ECL1i
- Aortoiliac Occlusive Disease Group (Active Comparator): Participants with non-aneurysmal aortoiliac occlusive disease, will be eligible for the study based on lifestyle limiting claudication (lack of blood flow to muscles causing cramping), pain in the feet or toes at rest, and/or tissue loss (leg or foot ulcers that don't heal or gangrene) that requires aortofemoral bypass. The aortofemoral bypass is not part of this research study.
  Interventions: Diagnostic Test: Aortoiliac Occlusive Disease Group - PET-CT imaging with injection of 64Cu-DOTA-ECL1i

INTERVENTIONS:
Diagnostic Test: Aortoiliac Occlusive Disease Group - PET-CT imaging with injection of 64Cu-DOTA-ECL1i — Patients from both genders, all ethnic groups, and between the ages of 45 and 75 will be considered for recruitment. We will recruit patients who have evidence of abdominal aortic aneurysm (AAA) as our study patient cohort. Patients with non-aneurysmal, atherosclerotic aortoiliac occlusive disease (n=3) will be enrolled in Aim 2A and undergo Cu-64 DOTA-ECL1i PET/CT.
  Arms: Aortoiliac Occlusive Disease Group
Diagnostic Test: AAA Group- PET-CT imaging with injection of 64Cu-DOTA-ECL1i — Patients from both genders, all ethnic groups, and between the ages of 45 and 75 will be considered for recruitment. We will recruit patients who have evidence of abdominal aortic aneurysm (AAA) as our study patient cohort. Patients with Abdominal aortic aneurysm (AAA) (n=5) will be enrolled in Aim 2B and undergo Cu-64 DOTA-ECL1i PET/CT and contrast-enhanced CT angiography between 7-14 days of their scheduled elective open repair surgery.
  Arms: AAA Group

SUMMARY:
The purpose of this research study is to look at whether an investigational imaging agent, 64Cu-DOTA-ECL1i, used during Positron Emission Tomography (PET)/ Computed Tomography (CT) scanning, can help to identify conditions that place patients at an increased risk for AAA rupture. The study is also looking more closely at cellular, molecular and inflammatory properties of the aortic wall. Having the ability to identify markers that predict AAA progression/expansion and risk for rupture could allow the physician to manage patients in a more individualized, personal way.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is a life-threatening degenerative vascular disease characterized by transmural aortic macrophage infiltration, elastin degradation, and reduction of smooth muscle cell content. AAAs occurs later in life and are especially prevalent in men over the age of 65. Patients typically remain asymptomatic until rupture, which is associated with high mortality. Currently, surgical repair is the only approach for AAA treatment, and there is no pharmacological intervention. Clinically, ultrasound and computed tomography measurement of aneurysm diameter represents the mainstay of management and the principal determinant of timing for elective surgical repair. However, this anatomy-based approach fails to provide useful information about the cellular and molecular processes associated with aneurysm expansion and rupture. Therefore, developing translatable molecular biomarkers, specifically expressed by aneurysms, is necessary to determine associated status and progression, capture the risk of rupture, and deliver personalized treatment.

ELIGIBILITY:
Non-Aneurysmal Patients, (Aim 2A, n=3)

Inclusion Criteria:

- Patients with aortoiliac occlusive disease causing lifestyle limiting claudication, rest pain, and/or tissue loss that requires aortofemoral bypass

Exclusion Criteria:

- Patients with aortoiliac occlusive disease, we will apply the same exclusion criteria as AAA patients.

Abdominal Aortic Aneurysm (AAA) Patients, (Aim 2B, n=5)

Inclusion Criteria:

* We will recruit asymptomatic patients with known AAAs by ultrasound, Doppler, and CT (men ≥ 5.5 cm, women ≥ 5.0cm);
* Both men and women, between the ages of 45 -75;
* With or without active tobacco use;

Exclusion Criteria:

* Inability to receive and sign informed consent;
* Has a history of hypersensitivity to contrast agent, Iopamidol (Isovue)
* Patients with Stage ≥ 4 chronic renal failure (calculated by modification of diet in renal disease eGFR equation [to minimize confounding imaging variables]);
* Inability to tolerate 60 minutes in a supine position with arms down at sides, as necessary for PET/CT;
* Severe claustrophobia;
* Positive pregnancy test or lactating;
* Has a history of hypersensitivity to 64Cu-DOTA-ECL1i or any of its excipients;
* Any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with collection of the data such as: Symptomatic/recently treated coronary disease, cancer requiring oncologic management, or autoimmune/inflammatory diseases (e.g., rheumatoid arthritis or multiple sclerosis) that are known to have increased associated expression of CCR2.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
First in-person CCR2 molecular imaging using 64Cu-DOTA-ECL1i PET/CT in AAA patient | 1-2 weeks
  Determine the background retention of 64Cu-DOTA-ECL1i in the abdominal aorta of patients with non-aneurysmal, atherosclerotic occlusive disease.
Perform 64Cu-DOTA-ECL1i PET/CT in AAA patients and correlate imaging readouts with tissue inflammatory biomarkers in patients undergoing open repair | 1-2 weeks prior to surgery
  Patients undergoing open AAA repair will be scheduled for PET/CT imaging at 1-2 weeks prior to surgery. This will be first-in-patient molecular imaging using CCR2 targeted 64Cu-DOTA-ECL1i in AAA patients undergoing open repair. The surgically removed aneurysmal tissue will be collected and processed for a complete characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Zayed, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No